CLINICAL TRIAL: NCT04462744
Title: Effectiveness of an Oral Health Educational Program on the Knowledge and Self-reported Practice of Primary School Teachers in Beni-Suef Towards Traumatic Dental Injuries: Before and After Study
Brief Title: the Effect of Educational Program on Teachers' Knowledge Self-reported Practice Towards TDIs
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Somaia Ahmed Mustafa, Bachelor degree 2014, Cairo University
Other Study IDs: teachers' knowledge of TDIs
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Dental Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: educational program — an oral health educational program regarding the emergency management of traumatic dental injuries.

SUMMARY:
The study aims at evaluating the effect of an oral health educational program on the knowledge and self-reported protocol of primary school teachers in Beni-Suef towards traumatic dental injuries.

DETAILED DESCRIPTION:
Traumatic dental injuries (TDIs) are considered a public health concern representing 5% of all injuries. According to the world health organization (WHO) about 16-40% of children across the world are subjected to TDIs with the most susceptible age group between 6-12 years old. Dental trauma may be caused by falls, blows to the face and sports which could be mild as concussion or subluxation, or complicated as avulsion ). The majority of the injuries took place at home followed by school, so teachers are one of the first to be present at the site of action, making their knowledge of emergency management essential to the provision of proper care to an injured child .

For example, in cases of avulsion of permanent tooth the proper management is to find the missing tooth and immediately replant, or transport the tooth in suitable transportation media, then referral to the dentist for treatment and follow up. The prognosis of such case mainly depends on the time between the injury and the replantation and the media of transportation . The unnecessary negative consequences of not providing proper first aid management in such case could lead to more time consuming and costly treatment and in a worst-case scenario permanent loss of one or more tooth . This could cause pain and have significant functional, esthetic, speech, and psychological effects on children thus affecting their quality of life .

A number of studies have evaluated the knowledge level of schoolteachers with respect to dental trauma and its emergency management concluded that teachers lack knowledge towards traumatic dental injuries. They recommended establishing oral health educational programs to raise the teachers' knowledge and improve their attitude towards TDIs . Other educational studies showed remarkable increase knowledge after oral health educational program and that is why educational programs and training are needed to improve proper management of traumatic injuries by schoolteachers and avoid unnecessary negative consequences.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females teachers.
* All ages and different periods of experience.
* From both private and public schools.
* Teachers in Beni-Suef district

Exclusion Criteria:

* Primary school teachers who refuse to participate.
* Teachers who attended any previous first aid course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary school teachers in Beni-Suef district of Beni-Suef governorate will be enrolled if they accept and are willing to participate.
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
The knowledge of primary school teachers regarding emergency management of traumatic dental injuries before and after an oral health educational program. | 2 months
  Previously validated self-administrated close ended questionnaire. the measuring unit eill be Percentage % Multiple choice question in the questionnaire.

SECONDARY OUTCOMES:
The self-reported practice of primary school teachers regarding emergency management of traumatic dental injuries before and after an oral health educational program. | 2 months
  Previously validated self-administrated close ended questionnaire. the outcome measuring unit will be Percentage % Multiple choice question in the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ola M Omar, professor, Study Chair — Cairo University
Locations (1):
- The district management of sducation, Banī Suwayf, Beni Suweif Governorate, Egypt